CLINICAL TRIAL: NCT03870269
Title: Using Virtual Reality (VR) Models for Robotic Prostatectomy - UNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceevra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-0904RP
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention Arm (Experimental): Subjects whose surgeon will be viewing VR models in addition to the source CT/MR image in connection with the case.
  Interventions: Device: Ceevra Reveal
- Control Arm (No Intervention): Subjects whose surgeon will only be viewing CT/MR images in connection with the case.

INTERVENTIONS:
Device: Ceevra Reveal — VR models generated using Ceevra Reveal are viewed by surgeons in connection with the case in addition to source CT/MR image.
  Arms: Intervention Arm

SUMMARY:
A prospective, randomized, controlled study designed to assess whether digital virtual reality (VR) models, created from existing CT scans and MRIs, provide surgeons with an improved understanding of their patients' anatomy, resulting in more efficient operations (robotic prostatectomy) and improved patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing robotic prostatectomy being performed by participating surgeon
* Patient is willing to be randomized between intervention and control arms

Exclusion Criteria:

* Patients with prior pelvic radiation
* Patients with prior androgen deprivation therapy
* Patients with prior localized ablative therapy
* Patients with prior TURP or other surgical BPH treatment

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Total operative time | During procedure, not to exceed 12 hours

SECONDARY OUTCOMES:
Blood loss (measured in cubic centimeters) | Measured at end of procedure, not to exceed 12 hours
Intraoperative conversion from robotic assisted laparoscopic procedure to open procedure | During procedure, not to exceed 12 hours
Intraoperative complication | During procedure, not to exceed 12 hours
Patient hospital stay | Measured at time of patient discharge, up to 10 days
Positive tumor margin (assessed via standard post-operative biopsy) | Measured 1-2 weeks after discharge
Postoperative Gleason Score | Measured up to 3 months after discharge
Postoperative oncologic stage (T stage) | Measured up to 3 months after discharge
Readmission | Measured up to 6 months after discharge
Postoperative prostate-specific antigen (PSA) | Measured up to 12 months after disccharge
Postoperative erectile function | Measured via survey up to 18 months after discharge
Postoperative continence | Measured via survey up to 18 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wallen, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided